CLINICAL TRIAL: NCT01554293
Title: A Randomized, Double-Blind, Placebo-Controlled Phase I Study To Determine The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Single Ascending Doses Of PBL 1427 In Healthy Volunteers
Brief Title: Study Of Single Ascending Doses Of PBL 1427 In Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Panacea Biotec Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PBL/CR/2011/05/CT
Record Dates: First submitted 2012-02-17; First posted 2012-03-14 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PBL 1427 capsules (Experimental)
  Interventions: Drug: PBL 1427 capsules
- Matching placebo (Placebo Comparator)
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Matching placebo — Matching Placebo, single dose
  Arms: Matching placebo
Drug: PBL 1427 capsules — PBL 1427 capsules 20 mg and 150 mg, single dose
  Arms: PBL 1427 capsules

SUMMARY:
PBL 1427 is a Dipeptidyl peptidase (DPP)-IV inhibitor being developed for treatment of type 2 diabetes. Although a number of DPP-IV inhibitors have been described, there still exists a need for new DPP-IV inhibitors that have better half-life, advantageous potency, stability and selectivity, less toxicity and/or better pharmacodynamic properties.

DETAILED DESCRIPTION:
As per the randomization schedule, capsule(s) of A or B will be administered to each subject with 240 mL of water at ambient temperature. Subjects will be instructed not to chew or crush the capsule(s) but to consume it as a whole. Compliance for dosing will be assessed by a thorough check of the oral cavity immediately after dosing. Administration of investigational products will be carried out while the subjects are in sitting posture and they will be instructed to remain seated for two hours after dosing except when clinically indicated to change the posture or in case of any natural exigency. Thereafter, the subjects will be allowed to engage in normal activities while avoiding severe physical exertion.

The following treatments in the below cohorts will be followed as given below:

Cohort 1: A single oral dose of 20 mg of PBL 1427 (n=6) or placebo (n=2) Cohort 2: A single oral dose of 40 mg (20 mg X 2 capsules) of PBL 1427 (n=6) or placebo (n=2) Cohort 3: A single oral dose of 80 mg (20 mg X 4 capsules) of PBL 1427 (n=6) or placebo (n=2) Cohort 4: A single oral dose of 150 mg of PBL 1427 (n=6) or placebo (n=2) Cohort 5: A single oral dose of 300 mg (150 mg X 2 capsules) of PBL 1427 (n=6) or placebo (n=2) Cohort 6: A single oral dose of 600 mg (150 mg X 4 capsules) of PBL 1427 (n=6) or placebo (n=2)

Dose levels may be modified and intermediate dose levels might be tested to determine the maximum tolerated dose (MTD)

The number of cohorts, dose levels, frequency and conditions of administration for the subsequent cohort may be altered by the Principal investigator and Sponsor after evaluation of the results of the previous group.

ELIGIBILITY:
Inclusion Criteria: Subjects to be enrolled in this trial must fulfil all of these criteria:

* Sex: male
* Age: 18-60 yr old, both inclusive
* Having a Body Mass Index (BMI) between 18.5-28 kg / m2 (both inclusive) and body weight not less than 45 kg
* Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; and to comply with the requirements of the entire study
* Voluntarily given written informed consent to participate in this study
* Be of normal health as determined by the principal investigator from medical history, physical examination and laboratory investigations, 12- lead ECG and X-ray chest of the subjects performed within 10 days prior to the admission of the study
* Ability and willingness to abstain from alcohol, methylxanthine-containing beverages or food (coffee, tea, coke, chocolate, "power drinks") and grapefruit (juice) from 48 h prior to each admission until study completion

Exclusion Criteria: Subjects meeting any of these criteria will not be enrolled in the study:

* Employees of FCRL or PBL
* Not willing to use contraceptives (preferably condoms) during sexual activity for the period of 3 months from the date of check-in
* History of hypersensitivity and / or intolerance to Dipeptidyl peptidase (DPP)-IV inhibitors or any other related compounds.
* History of anaphylaxis to drugs or allergic reactions in general, which the Investigator considers may affect the outcome of the study.
* Clinically abnormal ECG and Chest X-ray.
* Physical findings: clinically relevant abnormal physical findings (including body temperature) suggesting underlying pathologies or those which could interfere with the objectives of the study.
* Gastrointestinal disorders likely to influence drug absorption including acute gastrointestinal symptoms (e.g. nausea, vomiting, diarrhoea, heart burn), preceding one week to admission.
* Laboratory values that are significantly different than the normal reference range and/or are deemed to be of clinical significance by the investigator
* Presence of reactive disease markers of HIV 1 and II, HBsAg,, HCV or VDRL.
* Positive for alcohol breath test and/or urine drug screen (barbiturates, benzodiazepines, amphetamine, cocaine, opiates, tetra-hydro cannabinol).
* Any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
* History of Diabetes Mellitus or intake of any anti-diabetic medication
* Diseases: relevant history of renal, hepatic, cardiovascular, respiratory, skin, haematological, endocrine, neurological or gastrointestinal diseases. History of depression, psychosis, schizophrenia or any other severe psychiatric diseases, or epilepsy, or any other illness that may interfere with the aim of the study. History of any significant illness in the 4 weeks preceding the screening
* Medications: history of intake of any medications including over the counter medications (OTC) during the 4 weeks period prior to dosing with the IMP.
* Investigational drug trials: participation in the evaluation of any drug in the 3 months prior to the start of the study (dosing with IMP).
* Blood donation: Subjects who, through completion of this study, would have donated and/or lost more than 300 mL of blood in the past 12 weeks

Note: In case the blood loss is ≤ 200 mL; subject may be dosed 60 days after blood donation or last sample of the previous study

* Regular smokers who smoke more than 10 cigarettes daily or have difficulty abstaining from smoking for the duration of each study period.
* History of drug dependence or alcoholics

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with adverse events | Pre-dose and upto Day 5-9
  Safety and tolerability of PBL 1427 will be assessed after single ascending doses when administered alone on the basis of AEs, vital signs (BP, pulse rate, and body temperature), ECG, laboratory parameters and clinical assessment.
Pharmacokinetics Variables (Cmax, tmax, AUC, t1/2, kel, CL/F & Vz/F) | 48 hrs post dose
  Pharmacokinetic parameters of single ascending doses of PBL 1427 : For each subject, blood will be collected at the following time points: pre-dose, 0.25, 0.50, 0.75 1, 1.5, 2, 3, 4, 6, 8, 10, 14, 16, 20, 24, 36 and 48 h post-dose.

SECONDARY OUTCOMES:
Pharmacodynamics assessment (glucose, insulin, C-peptide, lactic acid) | Pre-dose and upto 4 h post-dose
  Pharmacodynamics will be assessed using markers like glucose, insulin, C-peptide, lactic acid and the exploratory markers plasma DPP-IV activity and plasma GLP-1 (Glucagon-like peptide I) levels
Exploratory markers (plasma DPP-IV activity and GLP-1 levels) | Pre-dose and upto 48 h after dosing
  Pharmacodynamics will be assessed using markers like glucose, insulin, C-peptide, lactic acid and the exploratory markers plasma DPP-IV activity and plasma GLP-1 (Glucagon-like peptide I) levels

CONTACTS AND LOCATIONS:
Overall Officials: Dr Deepak C Chilkoti, Principal Investigator — Head-Clinical Operations
Locations (1):
- Fortis Clinical Research Ltd, Faridabad, Haryana, India